CLINICAL TRIAL: NCT04400188
Title: A Phase Ⅰb/Ⅱ Study of Fluzoparib (SHR-3162) and Temozolomide With or Without SHR-1316 in Treating Patients With Replapsed Small Cell Lung Cancer
Brief Title: A Study of Fluzoparib (SHR-3162) and Temozolomide With or Without SHR-1316 in Treating Patients With Replapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3162-Ib-115
Record Dates: First submitted 2020-05-07; First posted 2020-05-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — fluzoparib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Fluzoparib (SHR-3162) combined with temozolomide or Fluzoparib (SHR-3162) and temozolomide with SHR-1316
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental A (part 1) : Fluzoparib + temozolomide (Experimental)
  Interventions: Drug: Fluzoparib; Drug: temozolomide
- Experimental B (part 2) : Fluzoparib + temozolomide + SHR-1316 (Experimental)
  Interventions: Drug: Fluzoparib; Drug: temozolomide; Biological: SHR-1316

INTERVENTIONS:
Drug: Fluzoparib — Given PO
Drug: temozolomide — Given PO
Biological: SHR-1316 — Given injection
  Arms: Experimental B (part 2) : Fluzoparib + temozolomide + SHR-1316

SUMMARY:
This research study is a multicentre phase Ⅰb/Ⅱ Study to evaluate the efficacy and safety of the combination of Fluzoparib (SHR-3162) and temozolomide with or without SHR-1316 in small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have recurrent small cell lung cancer confirmed by histology or cytology.
2. Failed one prior line of platinum-based chemotherapy.
3. Subjects must have measurable disease, at least one lesion, by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria (within 28 days prior to administration of study treatment) ;
4. Freshly acquired samples or archived specimens within 12 months before randomization must be provided.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Participant must have a life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Active or untreated central nervous system (CNS) metastases.
2. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
3. History of autoimmune disease.
4. Positive test result for human immunodeficiency virus (HIV).
5. Active hepatitis B or hepatitis C.
6. Severe infections.
7. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment.
8. Significant cardiovascular disease.
9. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Phase Ⅰb: Number of Subjects Experienced Any Dose-Limiting Toxicity (DLT) over the DLT period. | At the end of Cycle1 (each cycle is 21 days )
Phase Ⅰb: Determination of Recommended Phase II dose (RP2D) of Escalating Dose of Fluzoparib and temozolomide with or without SHR-1316. | Up to approximately 2 Years
Phase Ⅱ: Progression Free Survival (PFS) at four months. | Up to approximately 2 Years
Phase Ⅱ: Progression Free Survival (PFS) as Assessed by the Investigator according to RECIST v1.1. | Up to approximately 2 Years
  Progression Free Survival, defined as the time from randomization to first assessment of disease progression or death, whichever is earlier.

SECONDARY OUTCOMES:
Objective Response Rate | up to approximately 2 Years
  Objective Response Rate, determined using RECIST v1.1 criteria, defined as best overall response (complete or partial response) across all assessment time points.
Duration of Response | Up to approximately 2 Years
  Duration of Response, determined using RECIST v1.1 criteria.
Disease Control Rate | Up to approximately 2 Years
  Disease Control Rate, determined using RECIST v1.1 criteria.
Time to Response | Up to approximately 2 Years
  Time to Response, defined as the time from randomization to PR or CR.
Overall survival and overall survival at 6 months, 9months and 12 months | Up to approximately 1 Year
  Overall survival is the time interval from the date of randomization to death due to any reason or lost of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China